CLINICAL TRIAL: NCT01806467
Title: Continuous Thermodilution, Transpulmonary Thermodilution and Pressure Recording Analytical Method for Cardiac Output Measurement During Hemodynamic Instability: a Prospective Clinical Study
Brief Title: Validation of a New Method to Measure Cardiac Output: Comparison With Thermodilution
Status: Completed | Type: Observational
Sponsor: Università Politecnica delle Marche (Other)
Responsible Party: Principal Investigator, Abele Donati, MD, Professor, Università Politecnica delle Marche
Other Study IDs: 210107
Record Dates: First submitted 2013-02-26; First posted 2013-03-07 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Hemodynamic Instability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- critically ill patients: patients admitted to the medical-surgical ICU
- post-cardiac surgical patients: patients admitted to the post-cardiac surgical ICU

SUMMARY:
Many mini-invasive devices to monitor cardiac output (CO) have been introduced and among them the Pressure Recording Analytical Method (PRAM). The aim of this study is to assess the agreement of PRAM with the intermittent transpulmonary thermodilution (ThD) and continuous pulmonary ThD in measuring CO in hemodynamically unstable patients.

DETAILED DESCRIPTION:
Hemodynamic monitoring is important in critically ill patients. It is often used to assess a cardiovascular derangements, to help diagnosing the causes and to monitor the response to therapy.

Pulmonary thermodilution (ThD) is still considered the gold standard reference method for cardiac output (CO) measurement [1]. Its invasiveness, however, often limits or delays its application [2, 3]. In the last decades new less invasive hemodynamic monitoring systems have been developed. The majority of such new devices allows for continuous monitoring of CO and other hemodynamic variables [4].

Among the various less invasive techniques, the PiCCO (Pulse-induced Contour Cardiac Output) relies on the concept of the "pulse contour methodology" for providing beat-to-beat CO assessment. This method needs transpulmonary ThD calibration. This is a well validated dilution technique [5]. Another minimally invasive system is the Pressure Recording Analytical Method (PRAM). Unlike other systems with pulse contour analysis, the PRAM does not need external or internal calibration factors since it analyzes the pressure waveform at a frequency of 1000 Hz and computes the patient's cardiovascular system impedance using a mathematical algorithm based on the physical theory of perturbations. It only requires a connection to a femoral or radial artery catheter for the acquisition and analysis of the arterial pressure traces [6]. This new method has been validated under different experimental and clinical settings [6-9]. Limited data are available under conditions of hemodynamic instability [10-12]. So far, its accuracy and reliability in assessing CO in hemodynamically unstable patients needs yet to be clarified.

ELIGIBILITY:
Inclusion Criteria:

Hemodynamic instability in:

* septic shock
* pneumonia
* polytrauma
* chronic obstructive pulmonary disease
* heart failure
* post operative cardiosurgical patients

Exclusion Criteria:

* Atrial fibrillation
* Pacemaker or implantable cardiac defibrillator
* Aortic or mitral valve disease
* Intra-aortic balloon pump

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hemodynamic instability
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2011-08; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Blant-Altman test and coefficient of error of Cardiac Output measured with PRAM towards that measured with thermodilution | Study Period: 9 months
  Agreement between Cardiac Output measured with PRAM and cardiac output measured with thermodilution (both pulmonary and transpulmonary thermodilution) was determined by the Bland-Altman method. The precision of the measurements was given by the limits of agreement (LoA) (±1.96SD) of the mean difference of the methods compared. Upper and lower LoA were calculated as the bias ± 1.96SD. The percentage error was calculated as the LoA of the bias divided by the mean CO from two methods compared. Thirty per cent was considered an a priori criterion of interchangeability.

CONTACTS AND LOCATIONS:
Overall Officials: Abele Donati, MD, Principal Investigator — UPollitecnicaDM
Locations (1):
- AOU Ospedali Riuniti Ancona, Ancona, Ancona, Italy